CLINICAL TRIAL: NCT06580834
Title: Newborn Brain Test (NBT): Assessment of Newborn Brain Function Using Automated AI Assessment, Phase1 Feasibility Study
Brief Title: Newborn Brain Test (NBT)
Acronym: NBT
Status: Completed | Type: Observational
Sponsor: Professor Geraldine Boylan (Other)
Responsible Party: Sponsor-Investigator, Professor Geraldine Boylan, Professor, University College Cork
Organization: University College Cork (Other)
Other Study IDs: ECM 4 (tt) 05/12/2023
Record Dates: First submitted 2024-07-24; First posted 2024-08-30 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Seizures Newborn; Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonatal Intensive care Unit: 50% of the babies recruited will be from the Neonatal Intensive Care Unit. All term neonates ≥ 37 and ≤ 45 weeks corrected gestation age are eligible for the NBT study that do not have head trauma or broken skin on the scalp.
  Interventions: Device: Cergenx Wave
- Post Natal Ward: 50% of the babies recruited will be from the Post Natal Ward. All term neonates ≥ 37 and ≤ 45 weeks corrected gestation age are eligible for the NBT study that do not have head trauma or broken skin on the scalp.
  Interventions: Device: Cergenx Wave

INTERVENTIONS:
Device: Cergenx Wave — Short EEG recording using EEG amplifier with cloud based algorithm to assess brain injury.

SUMMARY:
The aim of the overall project is to develop the Newborn Brain Test (NBT), a novel platform to detect abnormal brain activity in infants at birth through an automated AI assessment. Easy to interpret results, provided in less than 15 minutes, will allow for immediate follow up by a medical team when abnormal brain function is detected.

NBT has been developed by INFANT's study partner CergenX (UCC Spinout company), who sponsors the study. INFANT is responsible for the clinical aspect of the project and will conduct a feasibility study of the device as well as a larger pivotal investigation.

DETAILED DESCRIPTION:
EEG activity will be recorded using the standard CE marked portable EEG amplifier with four electrodes on the scalp. The test will be controlled using a tablet. The captured waveforms will be sent to the cloud where the NBT Artificial Intelligence (AI) algorithm analyses EEG activity, analyses the data and decides whether the test was or was not completed successfully. The test takes approximately 15 minutes to complete. The device has been trained with EEG data from full term infants. It is not a diagnostic test, simply a screener.

The EEG and anonymised patient data collected during the NBT test will be processed and stored in the NBT secure AWS infrastructure. During the feasibility study, the result (EEG reading or result of AI algorithm) from the device will not be available to the research team so as not to influence clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* All neonates≥ 37 and ≤45 weeks gestational age
* Parental informed consent

Exclusion Criteria:

* Any Infant with head trauma or broken skin on the scalp
* Informed consent not obtained.

Ages: 37 Weeks to 45 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 90 babies will be recruited in total that meet the inclusion criteria above. 45 will be from the Neonatal Intensive care Unit and 45 from the Post natal Ward
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Assessing whether an acceptable EEG recording can be attained for the device on the first attempt for 80% of attempted recordings | Day 1
  Feasibility of the device is achieved if a good quality recording on the first attempt is achieved in at least 80% of infants , i.e. the device is not feasible if the success rate is <80%.
  Acceptable EEG in terms of technical quality for satisfactory review:
  * The recording should clearly be recording brain activity; if an electrode is poorly attached or detached, the EEG channel is likely to show continuous high amplitude/chaotic artifact which is not acceptable.
  * The brain activity for a term baby should contain continuous activity of mixed frequency content (delta, theta, alpha activity) with amplitudes ranging from 25-150µV.
  * The EEG should not be marred by persistent 50Hz due to high electrode impedance, that makes the recording unreadable.
  A 'majority' (50%+) of the EEG should be artefact free and readable.

SECONDARY OUTCOMES:
Time taken to complete assessment (as above) when a good quality recording is obtained for an infant on the first attempt | Day 1
  * A - Time taken to set up the device and put on the electrodes;
  * B - Time taken from electrode application to starting the device;
  * C - Time from pressing start on the device to results obtained;
  * D - Time from results obtained to removal of electrodes
  * Total time as above (A+B+C+D)
Time taken to complete assessment (as above) when a good quality recording is NOT obtained for an infant on the first attempt. | Day 1
  * A - Time taken to set up the device and put on the electrodes;
  * B - Time taken from electrode application to starting the device;
  * C - Time from pressing start on the device to results obtained;
  * D - Time from results obtained to removal of electrodes
  * Total time as above (A+B+C+D)
Number of attempts by a user before a good quality recording is achieved (Max 3 attempts) | Day 1
  A count of the failed attempts to make a recording. A failed recording is where no results are obtained from the tablet
Assessment of healthcare satisfaction with useability of the device and procedure derived from data captured during recordings and interviews. | The interviews will be conducted with the researchers after 10 weeks, after 20 weeks and at the end of the study - up to 30 weeks
  Information on healthcare professional satisfaction with the device will be collected by means of completed System Useability Scale (SUS) Questionnaires. Interviews will also be conducted with the healthcare professionals using pre-defined questions to gain further knowledge and information on the use of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Boylan, Professor, Study Director — University College Cork INFANT Centre
Locations (1):
- Cork University Maternity Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided